CLINICAL TRIAL: NCT03703089
Title: Gemcitabine and Nab-Paclitaxel in Pancreatic Adenocarcinoma With Positive Peritoneal Cytology as a Sole Metastatic Site, a Pilot Study
Brief Title: Gemcitabine & Nab-Paclitaxel in Pancreatic Adenocarcinoma With Positive Peritoneal Cytology
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP17130
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Positive Peritoneal Cytology
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine and Nab-Paclitaxel (Experimental): Participants received albumin-bound paclitaxel 125 mg/m^2 followed by gemcitabine 1000 mg/m^2 by intravenous infusion (IV) on Days 1, 8 and 15 of each 28 day cycle.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Administered by intravenous infusion over 30 minutes.
  Other Names: GEMZAR
Drug: nab-paclitaxel — Administered by intravenous infusion over 30-40 minutes.
  Other Names: Abraxane

SUMMARY:
Using gemcitabine and nab-paclitaxel, the investigators hope to establish the differential ability of local and cytologically positive disease to respond to this regimen, and in particular, the frequency of cytologic conversion from positive to negative in such patients. The investigators also can begin to assess the value of maximum local therapy, including surgery, in patients who cytologically convert from positive to negative.

DETAILED DESCRIPTION:
This research study is a Phase Ib clinical trial. It will assess the frequency of cytological conversion in patients with pancreatic adenocarcinoma and positive peritoneal cytology as a sole metastatic site following gemcitabine nab-paclitaxel.

Subjects must have a newly diagnosed stage 4 untreated metastatic pancreatic ductal cancer with positive peritoneal cytology as a sole metastatic site and meet all inclusion/exclusion criteria.

Treatment consists of 4 week treatment cycles. Nab-paclitaxel and gemcitabine will be administered on days 1,8, and 15.

ELIGIBILITY:
Inclusion Criteria:

1. Male, or a non-pregnant and non-lactating female.
2. Age ≥ 18 years.
3. Histologically proven diagnosis of pancreatic ductal adenocarcinoma (PDAC).
4. Radiographic and pathologic staging (including staging laparoscopy with peritoneal wash) consistent with pancreatic cancer, resectable, borderline resectable, or locally advanced or unresectable as defined by NCCN guidelines (http://www.nccn.org/professionals/physician_gls/f_guidelines.asp).
5. Laparoscopic confirmation that the PDAC is localized except for positive peritoneal cytology. Biliary stents are permitted.
6. Elevated CA19-9.
7. Measurable disease as defined by RECIST 1.1.
8. ECOG performance status of ≤ 1 (see Appendix A).
9. Adequate bone marrow reserves as evidenced by:

   * ANC ≥1,500 cells/μl; and
   * Platelet count ≥100,000 cells/μl; and
   * Hemoglobin ≥9 g/dL
10. Adequate hepatic function as evidenced by:

    * Serum total bilirubin 1.5 ≤; and
    * AST and ALT ≤2.5 x ULN; and
    * Alkaline phosphatase ≤2.5 x ULN
11. Adequate renal function as evidenced by creatinine ≤1.5 x ULN.
12. Women of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

    1. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption for 28 days prior to starting gemcitabine/nab- paclitaxel (including dose interruptions) and for 3 months after last dose of gemcitabine/nab-paclitaxel and
    2. Have a negative pregnancy test result at screening and agree to ongoing pregnancy testing at the Investigator's discretion during the course of the study. This applies even if the subject practices true abstinence from heterosexual contact.
13. Male subjects must practice true abstinence or agree to use a condom during sexual contact with a female of childbearing potential or a pregnant female while on treatment (including during dose interruptions) with gemcitabine/nab-paclitaxel and for 3 months following the last dose of gemcitabine/nab- paclitaxel, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Prior chemotherapy or radiation for pancreatic cancer.
2. CA19-9 non-expressing.
3. Previous (within the past 5 years) or concurrent, malignancy diagnosis, except non-melanoma skin cancer and in situ carcinomas.
4. History of allergy or hypersensitivity to human, humanized or chimeric monoclonal antibodies.
5. Any medical or surgical condition that may place the subject at increased risk while on study.
6. Any condition potentially decreasing compliance to study procedures.
7. Participation in any other clinical protocol or investigational trials within 60 days prior to Day 1, Cycle 1.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Current abuse of alcohol or illicit drugs.
10. Any medical condition that, in the opinion of the Investigator, may pose a safety risk to the subject, may confound the assessment of safety and efficacy, or may interfere with study participation.
11. Have ≥ Grade 2 pre-existing peripheral neuropathy (per CTCAE).
12. Inability or unwillingness to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of cytological conversion | An average of 6 months
  To assess the frequency of cytological conversion in patients with pancreatic adenocarcinoma and positive peritoneal cytology as a sole metastatic site following gemcitabine nab-paclitaxel.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  Assess progression-free survival (PFS)
Overall survival (OS) | Up to 5 years
  Assess overall survival (OS).
Overall response rate | Up to 5 years
  Assess overall response rate.
Response rate by CA19-9 | An average of 1 year
  Assess response rate as measured by serial CA19-9 determinations.
Response rate by RECIST criteria 1.1 | Assessment approximately every 8 weeks during treatment up to 5 years
  Assess response rate as measured by RECIST criteria 1.1 radiographic criteria.
Ability to achieve R0 (complete) | At time of surgery, approximately 6 months after enrollment
  Assess the ability to achieve R0 (complete) resection rate in anatomically appropriate patients.
Local disease control rate. | Baseline, and approximately every 8 weeks during treatment. Up to 5 years
  Measure the local disease control rate.
Pattern of disease recurrence | Up to 5 years
  Observe the pattern of disease recurrence (both in anatomic space and time) in the above patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent J Picozzi, MD, Principal Investigator — Virginia mason medical Center
Locations (1):
- Virginia mason medical Center, Seattle, Washington, United States